CLINICAL TRIAL: NCT02529501
Title: Factors Influencing the Choice of Anesthesia (Spinal Anesthesia or Short General Anesthesia) in Outpatient Surgery
Brief Title: Spinal Versus General Anesthesia for Ambulatory Anesthesia
Acronym: BAG
Status: Completed | Type: Observational
Sponsor: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: BAG
Record Dates: First submitted 2015-07-27; First posted 2015-08-20 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-05

CONDITIONS: Spinal Anesthesia; Short General Anesthesia; Outpatient Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SA: Patients undergoing spinal anesthesia
- GA: Patients undergoing short general anesthesia

SUMMARY:
The purpose of this study is to describe, in real-life conditions, the factors influencing the choice of anesthesia (spinal anesthesia or short general anesthesia) in outpatient surgery.

DETAILED DESCRIPTION:
This is a cross-sectional, observational, prospective, multicentre study, conduct in France among a representative sample of anesthesiologists.

The factors influencing the choice of anesthesia (spinal anesthesia or short general anesthesia) will be assessed in patients undergoing an outpatient surgery. Data will be collected by the physician during the inclusion visit (peripostoperative consultation). Additional data regarding the patient's perception (pain and satisfaction) will be collected using a self-questionnaire 7 days after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing an ambulatory surgery
* Patients for whom either a spinal anesthesia or a short general anesthesia is planned
* Patients accepting and able to complete a self-administered questionnaire in French language
* Informed patients who accept the computer processing of their medical data and their right of access and correction

Exclusion Criteria:

* Patients with contra-indications to elective ambulatory surgery
* Emergency surgeries
* Patient for which both spinal anesthesia and short general anesthesia coexist
* Patients with contra-indications to spinal anesthesia (due to surgical procedure site, comorbidities or patient's treatment)
* Patients participating or having participated in the previous month in a clinical trial in anaesthesiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery under spinal anesthesia or short general anesthesia will be informed about the study and will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 595 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Factors influencing the choice of anesthesia (spinal anesthesia or short general anesthesia | During the perioperative consultation (patients are included at the time of the perioperative consultation prior to their surgery): baseline visit
  All proposed factors will be described using a 4-levels verbal scale (decisive / important / of little importance / unimportant). The factors will be described from the questionnaire completed by the investigator during the inclusion visit, before the surgery.
  Decisive factors for the choice of anesthesia will be described and compared between the two subgroups.spinal anesthesia and short general anesthesia.

SECONDARY OUTCOMES:
Patients' characteristics in each subgroups | At the time of the perioperative consultation prior to their surgery (start of the inclusion visit or baseline visit)
  Patients' characteristics (demographic data, ASA physical status, risk factors...) will be described from the questionnaire completed by the investigator during the inclusion visit, before the surgery.
Postoperative period from waking up to eligibility for discharge from hospital according to the type of anesthesia | Up to 24h after the surgery
  Will be described from the questionnaire completed by the investigator during the inclusion visit, after the surgery.
Patients' satisfaction according to the type of anesthesia based on 2 questions using a 4-levels verbal scale | 7 days after surgery (i.e. 7 days after the inclusion)
  Will be described from the self-questionnaire completed by the patient 7 days after the surgery.
Patients' pain according to the type of anesthesia using a VAS scale | Up to 7 days after surgery
  Will be described from the self-questionnaire completed by the patient 7 days after the surgery.
Costs of spinal and general anesthesia | The day of the surgery
  Will be described from the questionnaire completed by the investigator during the inclusion visit.
Use and safety of Baritekal® (prilocaine) if applicable | During surgery
  Modalities of spinal anesthesia with prilocaine. Percentage and nature of adverse effect (serious or not) after intrathecal anaesthesia with prilocaine.

CONTACTS AND LOCATIONS:
Overall Officials: Hélène HERMAN-DEMARS, MD, Study Director — Nordic Pharma
Locations (1):
- Nordic Pharma, Paris, France

REFERENCES:
- [Derived] Capdevila X, Aveline C, Delaunay L, Bouaziz H, Zetlaoui P, Choquet O, Jouffroy L, Herman-Demars H, Bonnet F. Factors Determining the Choice of Spinal Versus General Anesthesia in Patients Undergoing Ambulatory Surgery: Results of a Multicenter Observational Study. Adv Ther. 2020 Jan;37(1):527-540. doi: 10.1007/s12325-019-01171-6. Epub 2019 Dec 11. PMID 31828612